CLINICAL TRIAL: NCT00141102
Title: Double-Blind, Triple Dummy, Parallel-Group, Randomized, Six-Month Study To Compare Celecoxib (200 Mg BID) With Diclofenac Sr (75 Mg BID) Plus Omeprazole (20 Mg QD) For Gastrointestinal Events In Subjects With Osteoarthritis And Rheumatoid Arthritis At High-Risk Of Gastrointestinal Adverse Events
Brief Title: Study Of Celecoxib Or Diclofenac And Omeprazole For Gastrointestinal (GI) Safety In High GI Risk Patients With Arthritis
Acronym: CONDOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3191084
Record Dates: First submitted 2005-08-29; First posted 2005-09-01 (Estimated); Results first posted 2010-06-11 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid
Keywords: GI events in high risk GI arthritis patients
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid | interventions — Celecoxib; Diclofenac; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Active Comparator)
  Interventions: Drug: Diclofenac + Omeprazole

INTERVENTIONS:
Drug: Celecoxib — Participants are assigned to one of two groups in parallel for the duration of the study
  Arms: A
Drug: Diclofenac + Omeprazole — Participants are assigned to one of two groups in parallel for the duration of the study
  Arms: B

SUMMARY:
To determine whether celecoxib is superior to combined therapy with diclofenac and omeprazole in the incidence of clinically significant upper and/or lower gastrointestinal (GI) events in high GI risk subjects with osteoarthritis and/or rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of OA or RA and who are expected to require regular anti-inflammatory therapy for arthritis symptom management
* Subjects must be aged 60 years or older with or without a history of gastroduodenal (GD) ulceration; or be of any age 18 years or older and have had documented evidence of GD ulceration 90 days or more prior to the screening visit

Exclusion Criteria:

* Active GD ulceration or GD ulceration within 90 days of the screening visit.
* Concomitant use of low dose aspirin
* Previous MI, stroke or significant vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4484 (Actual)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (144):
- Belgium (4):
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Liège
- Brazil (5):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (8):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Ste Foy, Quebec
- China (6):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Chengdu, Sichuan
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Tianjin
- Colombia (4):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Floridablanca, Santander Department
- Costa Rica (3):
  - Pfizer Investigational Site, Cartago
  - Pfizer Investigational Site, Heredia
  - Pfizer Investigational Site, San José
- Croatia (2):
  - Pfizer Investigational Site, Opatija
  - Pfizer Investigational Site, Zagreb
- Czechia (5):
  - Pfizer Investigational Site, Pilsen, Bory
  - Pfizer Investigational Site, Ostrava, Trebovice
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
- Ecuador (3):
  - Pfizer Investigational Site, Cuenca, Azuay
  - Pfizer Investigational Site, Guayaquil, Guayas
  - Pfizer Investigational Site, Quito, Pichincha
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- France (2):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Dijon
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Deggingen
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hoyerswerda
  - Pfizer Investigational Site, Künzing
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Nuremberg
- Pfizer Investigational Site, Thessaloniki, Greece
- Pfizer Investigational Site, Guatemala City, Guatemala
- Hong Kong (2):
  - Pfizer Investigational Site, Lai Chi Kok
  - Pfizer Investigational Site, Shatin
- India (3):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Ludhiana, Punjab
- Pfizer Investigational Site, Riga, Latvia
- Lithuania (4):
  - Pfizer Investigational Site, Alytus
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Klaipėda
  - Pfizer Investigational Site, Vilnius
- Netherlands (3):
  - Pfizer Investigational Site, Vlaardingen, South Holland
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Leidschendam
- Pfizer Investigational Site, Panama City, Panama
- Peru (2):
  - Pfizer Investigational Site, Surco, Lima region
  - Pfizer Investigational Site, Lima
- Portugal (3):
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Ponta Delgada
  - Pfizer Investigational Site, Ponte de Lima
- Russia (5):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Petrozavodsk
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
  - Pfizer Investigational Site, Yekaterinburg
- Serbia (3):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Niška Banja
  - Pfizer Investigational Site, Novi Sad
- Singapore (2):
  - Pfizer Investigational Site, Sinapore
  - Pfizer Investigational Site, Singapore
- South Africa (8):
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Parow, Western Cape
  - Pfizer Investigational Site, Bellville
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Kempton Park
  - Pfizer Investigational Site, Observatory Cape Town
- Pfizer Investigational Site, Seoul, South Korea
- Spain (8):
  - Pfizer Investigational Site, Partida de Bacarot, Alicante
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Barakaldo, Vizcaya
  - Pfizer Investigational Site, Ávila
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Zaragoza
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Norrköping
- Taiwan (5):
  - Pfizer Investigational Site, Kaohsiung Hsien
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District
- Ukraine (11):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Ivano-Frankivsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kiev
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lutsk
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Simferopol
  - Pfizer Investigational Site, Zaporizhzhia
- United Kingdom (25):
  - Pfizer Investigational Site, Helensburgh, Argyle & Clyde
  - Pfizer Investigational Site, Maidenhead, Berks
  - Pfizer Investigational Site, Aston Clinton, Buckinghamshire
  - Pfizer Investigational Site, St Austell, Cornwall
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Aldershot, Hampshire
  - Pfizer Investigational Site, Basingstoke, Hampshire
  - Pfizer Investigational Site, Odiham, Hampshire
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Harrow, Middlesex
  - Pfizer Investigational Site, Camberley, Surrey
  - Pfizer Investigational Site, East Horsley, Leatherhead, Surrey
  - Pfizer Investigational Site, Pound Hill, Crawley, WEST Sussex
  - Pfizer Investigational Site, Bradford-on-Avon, Wiltshire
  - Pfizer Investigational Site, Chippenham, Wiltshire
  - Pfizer Investigational Site, Upton, Wirral
  - Pfizer Investigational Site, Bexhill-on-Sea
  - Pfizer Investigational Site, Canterbury
  - Pfizer Investigational Site, Chesterfield
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Peterborough
  - Pfizer Investigational Site, Saint Leonards-on-Sea
  - Pfizer Investigational Site, Swindon
  - Pfizer Investigational Site, Vale of Glamorgan
  - Pfizer Investigational Site, Wansford

REFERENCES:
- [Derived] Kellner HL, Li C, Essex MN. Celecoxib and Diclofenac Plus Omeprazole are Similarly Effective in the Treatment of Arthritis in Patients at High GI Risk in the CONDOR Trial. Open Rheumatol J. 2013 Nov 13;7:96-100. doi: 10.2174/1874312901307010096. eCollection 2013. PMID 24358067
- [Derived] Chan FK, Lanas A, Scheiman J, Berger MF, Nguyen H, Goldstein JL. Celecoxib versus omeprazole and diclofenac in patients with osteoarthritis and rheumatoid arthritis (CONDOR): a randomised trial. Lancet. 2010 Jul 17;376(9736):173-9. doi: 10.1016/S0140-6736(10)60673-3. Epub 2010 Jun 16. PMID 20638563
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191084&StudyName=Study%20Of%20Celecoxib%20Or%20Diclofenac%20And%20Omeprazole%20For%20Gastrointestinal%20%28GI%29%20Safety%20In%20High%20GI%20Risk%20Patients%20With%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: 200 milligrams (mg) twice daily (BID) plus omeprazole placebo and diclofenac slow release (SR) placebo
- Oral Diclofenac Plus Omeprazole: Oral diclofenac SR (75 mg BID) plus omeprazole (20 mg once daily [QD]) and celecoxib placebo.
Period: Overall Study
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Started | 2238 | 2246
Received Treatment | 2223 | 2237
Completed | 1730 | 1621
Not Completed | 508 | 625
Not completed — Adverse Event | 233 | 305
Not completed — Laboratory Abnormality | 9 | 33
Not completed — Lack of Efficacy | 21 | 26
Not completed — Lost to Follow-up | 29 | 32
Not completed — Other | 87 | 76
Not completed — Withdrawal by Subject | 112 | 142
Not completed — Randomized But Did Not Receive Treatment | 15 | 9
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib: 200 mg BID plus omeprazole placebo and diclofenac SR placebo
- Oral Diclofenac Plus Omeprazole: Oral diclofenac SR (75 mg BID) plus omeprazole (20 mg QD) and celecoxib placebo.
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole | Total
Number analyzed (Participants) | 2238 | 2246 | 4484
Age, Customized [Number; unit: participants]
  < 55 years | 176 | 164 | 340
  55 to 59 years | 122 | 113 | 235
  60 to 64 years | 721 | 742 | 1463
  65 to 69 years | 623 | 618 | 1241
  70 to 74 years | 361 | 390 | 751
  > = 75 years | 235 | 219 | 454
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1848 | 1822 | 3670
  Male | 390 | 424 | 814

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinically Significant Upper and/or Lower Gastrointestinal Events (CSULGIEs)
Description: CSULGIE=any of the following: gastroduodenal (GD) hemorrhage; gastric outlet obstruction; GD, small or large bowel perforation; small or large bowel hemorrhage; clinically significant anemia of defined GI origin; acute GI hemorrhage of unknown origin, including presumed small bowel hemorrhage; clinically significant anemia of presumed occult GI origin including possible small bowel blood loss. Subjects were assessed by an independent GI Events Adjudication Committee, who were blinded to study treatment assignments.
Time Frame: 6 month treatment duration
Population: Intent-to-Treat (ITT) = included all randomized subjects. n = number of subjects with events confirmed by the committee.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2238 | 2246
participants | 20 | 81
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p < 0.0001, Life Table Extension; Stratified by history of GD ulceration and by region; Odds Ratio (OR) = 4.32

2. Secondary Outcome: Number of Subjects With CSULGIES or Symptomatic Ulcers (SUs)
Description: CSULGIE=any of the following: GD hemorrhage; gastric outlet obstruction; GD, small or large bowel perforation; small or large bowel hemorrhage; clinically significant anemia of defined GI origin; acute GI hemorrhage of unknown origin, including presumed small bowel hemorrhage; clinically significant anemia of presumed occult GI origin including possible small bowel blood loss. Subjects with evaluation at an event visit and found to have an ulcer on endoscopy, but did not meet any criteria considered for the primary endpoint by the GI committee were designated as having an SU.
Time Frame: 6 month treatment duration
Population: ITT. n = number of subjects with CSULGIEs or SUs as confirmed by the committee.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2238 | 2246
participants | 25 | 92
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p < 0.0001, Life Table Extension; Stratified by history of GD ulceration and by region; Odds Ratio (OR) = 3.93

3. Secondary Outcome: Change From Baseline in Patient's Global Arthritis Assessment at Month 6/Early Termination (ET)
Description: Subjects rated response to question: "Considering all the ways the osteoarthritis or rheumatoid arthritis affects you, how are you doing today?" using a 1 to 5 grading scale where 1=very good and 5=very poor.
Time Frame: Month 6/Early Termination (ET)
Population: ITT. Number of Participants Analyzed = number of subjects with data available for the analysis. Last Observation Carried Forward (LOCF) method was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2207 | 2213
scores on a scale | 0.754 (0.020) | 0.773 (0.019)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.4146, ANCOVA; Fixed effects of region and history of GD ulceration with Baseline covariate; Least Squares (LS) Mean Difference = -0.019, 95% CI 2-sided [-0.06 to 0.03], Standard Error of Mean 0.023

4. Secondary Outcome: Number of Subjects With SUs
Description: Subjects with evaluation at an event visit and found to have an ulcer on endoscopy, but did not meet any criteria considered for the primary endpoint by the GI committee were designated as having an SU.
Time Frame: 6 month treatment duration
Population: ITT.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2238 | 2246
participants | 5 | 11
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.1132, Life Table Extension; Stratified by history of GD ulceration and by region; Odds Ratio (OR) = 2.29

5. Secondary Outcome: Number of Subjects With CSULGIEs by History of GD Ulceration
Description: as for outcome 1
Time Frame: 6 month treatment duration
Population: ITT. n = number of subjects who had history or no history of GD ulceration.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2238 | 2246
participants
  History of GD Ulceration (n=395, 400) | 7 | 13
  No History of GD Ulceration (n=1843, 1846) | 13 | 68

6. Secondary Outcome: Number of Subjects With Moderate to Severe Abdominal Symptoms
Description: Abdominal symptoms were defined by the Medical Dictionary for Regulatory Activities MedDRA System Organ Class (SOC) 'Gastrointestinal Disorders' and keeping high level group term (HLGT) equal to "Gastrointestinal Signs and Symptoms".
Time Frame: 6 month treatment duration
Population: ITT
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2238 | 2246
participants | 132 | 162
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.0495, Life Table Extension; Stratified by history of GD ulceration and by region; Odds Ratio (OR) = 1.26

7. Secondary Outcome: Number of Subjects Withdrawn Due to GI Adverse Events (AEs)
Description: GI AEs were defined using MedDRA SOC "Gastrointestinal Disorders" but excluding the following HLGTs: Benign Neoplasms Gastrointestinal; Dental and Gingival Conditions; Oral Soft Tissue Conditions; Salivary Gland Conditions; and Tongue Conditions.
Time Frame: 6 month treatment duration
Population: ITT
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2238 | 2246
participants | 114 | 167
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.0006, Life Table Extension; Stratified by history of GD ulceration and by region; Odds Ratio (OR) = 1.52

8. Secondary Outcome: Change From Baseline in Hemoglobin at Month 6/ET
Time Frame: Month 6/ET
Population: Safety population = all randomized subjects who received at least 1 dose of study medication. Number of Participants Analyzed = number of subjects with analyzable data.
Measure: Least Squares Mean (Standard Error); unit: grams (g)/deciliter (dL)
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2184 | 2167
grams (g)/deciliter (dL) | -0.017 (0.019) | -0.423 (0.019)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Fixed effects of region and history of GD ulceration with Baseline covariate; LS Mean Difference = 0.406, 95% CI 2-sided [0.36 to 0.45], Standard Error of Mean 0.022

9. Secondary Outcome: Change From Baseline in Hematocrit at Month 6/ET
Time Frame: Month 6/ET
Population: Safety population. Number of Participants Analyzed = number of subjects with analyzable data.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2184 | 2167
percent | -0.306 (0.059) | -1.425 (0.059)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p < 0.0001, ANCOVA; Fixed effects of region and history of GD ulceration with Baseline covariate; LS Mean Difference = 1.118, 95% CI 2-sided [0.98 to 1.25], Standard Error of Mean 0.069

10. Secondary Outcome: Number of Subjects With a Clinically Significant Decrease From Baseline in Hematocrit and/or Hemoglobin
Description: A clinically significant decrease from baseline was defined as a fall in hematocrit > = 10 percentage points and/or hemoglobin > = 2 g/dL.
Time Frame: 6 month treatment duration
Population: Safety population. Number of Participants Analyzed = number of subjects with analyzable data.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2184 | 2167
participants | 45 | 123
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by history of GD ulceration and by region; Relative Risk = 2.748, 95% CI 2-sided [1.96 to 3.84]

11. Secondary Outcome: Number of Subjects With Hepatic AEs in Gamma Glutamyl-Transferase (GGT), Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) of 3 Times the Upper Limit of Normal (ULN)
Description: GGT ULN was 49 international units (IU)/liter (L) for females and 61 IU/L for males, AST ULN was 37 IU/L for females and 39 IU/L for males, and ALT ULN was 43 IU/L for females and 45 IU/L for males.
Time Frame: 6 month treatment duration
Population: Safety population. Number of participants analyzed = number of subjects with analyzable data.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2223 | 2237
participants
  GGT | 26 | 86
  AST | 8 | 12
  ALT | 13 | 27
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; GGT; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Relative Risk = 3.329, 95% CI 2-sided [2.156 to 5.141]
Statistical Analysis 2: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; AST; Test type: Superiority or Other; p = 0.3809, Fisher Exact; Relative Risk = 1.509, 95% CI 2-sided [0.618 to 3.684]
Statistical Analysis 3: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; ALT; Test type: Superiority or Other; p = 0.0264, Fisher Exact; Relative Risk = 2.089, 95% CI 2-sided [1.081 to 4.038]

12. Secondary Outcome: Change From Baseline in Hepatic Measures of GGT, AST or ALT to Month 6/ET
Time Frame: Month 6/ET
Population: Safety population. Number of participants analyzed = number of subjects with analyzable data.
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2223 | 2237
IU/L
  GGT | -2.689 (0.591) | 7.455 (0.592)
  AST | -0.901 (0.239) | 1.490 (0.239)
  ALT | -1.151 (0.364) | 5.213 (0.364)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; GGT; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -10.144, 95% CI 2-sided [-11.51 to -8.78], Standard Error of Mean 0.697
Statistical Analysis 2: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; AST; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -2.391, 95% CI 2-sided [-2.94 to -1.84], Standard Error of Mean 0.281
Statistical Analysis 3: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; ALT; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -6.364, 95% CI 2-sided [-7.20 to -5.52], Standard Error of Mean 0.428

13. Secondary Outcome: Change From Baseline in Iron Binding Capacity to Month 6/ET
Time Frame: Month 6/ET
Population: Safety population. Number of participants analyzed = number of subjects with analyzable data.
Measure: Least Squares Mean (Standard Error); unit: microgram (ug)/dL
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2185 | 2171
microgram (ug)/dL | 2.517 (1.158) | 1.952 (1.161)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.6795, ANCOVA; Fixed effects of region and history of GD ulceration with Baseline covariate; LS Mean Difference = 0.565, 95% CI 2-sided [-2.11 to 3.24], Standard Error of Mean 1.366

14. Secondary Outcome: Change From Baseline in Ferretin to Month 6/ET
Time Frame: Month 6/ET
Population: Safety population. Number of participants analyzed = number of subjects with analyzable data.
Measure: Least Squares Mean (Standard Error); unit: ug/dL
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2185 | 2170
ug/dL | -3.396 (2.224) | -1.990 (2.228)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.5920, ANCOVA; Fixed effects of region and history of GD ulceration with Baseline covariate; LS Mean Difference = -1.406, 95% CI 2-sided [-6.55 to 3.74], Standard Error of Mean 2.624

15. Secondary Outcome: Change From Baseline in C-Reactive Protein to Month 6/ET
Time Frame: Month 6/ET
Population: Safety population. Number of participants analyzed = number of subjects with analyzable data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2185 | 2171
mg/dL | 0.058 (0.032) | 0.073 (0.032)
Statistical Analysis 1: Comparison: Celecoxib vs Oral Diclofenac Plus Omeprazole; Test type: Superiority or Other; p = 0.6819, ANCOVA; Fixed effects of region and history of GD ulceration with Baseline covariate; LS Mean Difference = -0.015, 95% CI 2-sided [-0.09 to 0.06], Standard Error of Mean 0.038

16. Other Pre Specified Outcome: Number of Subjects Alive at the Post Trial Interview
Description: Interview occurred via telephone to obtain follow-up mortality and hospitalization information.
Time Frame: 6 months following last dose
Population: Safety population. Number of participants analyzed = number of subjects with follow-up information available.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2047 | 2048
participants | 2018 | 2023

17. Other Pre Specified Outcome: Number of Subjects Hospitalized in Last 6 Months at the Post Trial Interview
Description: Interview occurred via telephone to obtain follow-up mortality and hospitalization information.
Time Frame: 6 months following last dose
Population: Safety population. Number of participants analyzed = number of subjects with follow-up information available.
Measure: Number; unit: participants
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Number analyzed (Participants) | 2047 | 2048
participants | 82 | 79

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib | Oral Diclofenac Plus Omeprazole
Serious Adverse Events (participants affected / at risk) | 61/2223 | 61/2237
Other Adverse Events (participants affected / at risk) | 530/2223 | 669/2237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=2223) | Oral Diclofenac Plus Omeprazole (N=2237)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 2
Burn infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Eye burns (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 2
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Open reduction of fracture (Surgical and medical procedures) | 1 | 0
Prolapse repair (Surgical and medical procedures) | 1 | 0
Rectocele repair (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=2223) | Oral Diclofenac Plus Omeprazole (N=2237)
Abdominal pain upper (Gastrointestinal disorders) | 96 | 133
Diarrhoea (Gastrointestinal disorders) | 79 | 168
Dyspepsia (Gastrointestinal disorders) | 137 | 111
Gastritis (Gastrointestinal disorders) | 32 | 44
Nausea (Gastrointestinal disorders) | 33 | 66
Oedema peripheral (General disorders) | 46 | 67
Nasopharyngitis (Infections and infestations) | 55 | 46
Haemoglobin decreased (Investigations) | 27 | 72
Headache (Nervous system disorders) | 66 | 48
Hypertension (Vascular disorders) | 76 | 84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.